CLINICAL TRIAL: NCT06470542
Title: Two-level Erector Spinae vs iPack With ACB Plane Block in Total Knee Arthroplasty
Brief Title: Two-level ESPB in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9/2024
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPACK + ACB (Active Comparator): Ultrasound-guided iPACK +ACB
  Interventions: Drug: 2 x 20 ml of Ropivacaine 0.2% Injectable Solution
- Two-Level ESPB (Active Comparator): Bi-level Ultrasound-guided ESPB et the L1 and S1
  Interventions: Drug: 2 x 20ml of Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: 2 x 20 ml of Ropivacaine 0.2% Injectable Solution — 2 x 20ml 0.2% Ropivacaine - ultrasound-guided iPACK + ACB
  Other Names: iPACK + ACB
  Arms: iPACK + ACB
Drug: 2 x 20ml of Ropivacaine 0.2% Injectable Solution — 2 x 20ml 0.2% ropivacaine - ultrasound-guided ESPB at the L1 and S1 level
  Other Names: Erector spinae plane block (ESPB)
  Arms: Two-Level ESPB

SUMMARY:
Effect of two-level ESPB in Total Knee Arthroplasty

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopaedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prostheses. Regional anaesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total hip arthroplasty
* patients aged >65 and <100 years
* patients able to provide informed consent
* patients able to reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a language barrier

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption | 48 hours after surgery
  Total opioid consumption after surgery - within 48 hours after surgery

SECONDARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
NLR | 24 hours after surgery
  neutrophil-to-lymphocyte ratio
NLR | 48 hours after surgery
  neutrophil-to-lymphocyte ratio
PLR | 24 hours after surgery
  platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: Yes
Detailed data sharing plan to be defined
Time Frame: Data will be shared following the trial completion
Access Criteria: Eligible researchers